CLINICAL TRIAL: NCT07042724
Title: PerSonalized nuTrition and physicAl exeRcise Intervention to Enhance earLy-staGe NSCLC ouTcomes: the STARLighT Study
Brief Title: Exercise and Nutrition on Early-stage NSCLC Outcomes: the STARLighT Study
Acronym: STARLighT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universita di Verona (Other)
Responsible Party: Principal Investigator, Sara Pilotto, MD, Ph.D, Universita di Verona
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Prog. 577CET
Record Dates: First submitted 2025-06-09; First posted 2025-06-29 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Lung Cancer (NSCLC)
Keywords: physical exercise;; nutrition;; lung cancer;
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Motor Activity | interventions — Exercise; Diet Therapy; Nutritional Status

STUDY DESIGN:
Intervention Model Description: A master clinical protocol will be set up to evaluate the exercise and nutritional interventions in different cohorts of patients diagnosed with non-oncogene addicted with early-stage NSCLC.
  Cohort A, assessing exercise and nutrition in the neoadjuvant lung cancer setting, will exploit a single-arm design.
  Cohort B, assessing exercise and nutrition in the adjuvant lung cancer setting, will exploit a randomized controlled design.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cohort A - neoadiuvant setting - interventional arm (Experimental): This arm will include patients undergoing neoadjuvant chemoimmunotherapy. The administered intervention will consist of a combination of exercise and nutrition support for the entire neoadjuvant treatment period.
  Interventions: Behavioral: Physical exercise and nutrition intervention for the neoadjuvant setting
- Cohort B - adiuvant setting - interventional arm (Experimental): This arm will include patients undergoing adjuvant treatment as per standard of care. The administered intervention will consist of a combination of exercise and nutrition support lasting 6 months.
  Interventions: Behavioral: Physical exercise and nutrition for the adjuvant setting
- Cohort B - adiuvant setting (Active Comparator): This arm will include patients undergoing adjuvant treatment as per standard of care. The administered intervention, lasting 6 months, will consist of health educational materials, including the benefits of exercise and nutrition during cancer care, the current recommendations, and information on how to pursue them, as well as strategies to achieve and maintain a healthy psychological status
  Interventions: Behavioral: Health educational material

INTERVENTIONS:
Behavioral: Physical exercise and nutrition intervention for the neoadjuvant setting — * Physical exercise: 3 sessions/week. It will comprise high-intensity interval training consisting of 2 minutes of high-intensity intervals interspersed with 2 minutes of active recovery completed at mild intensity. The number of intervals will start with five and progress based on the patient's exercise response. Resistance training will include 3-4 exercises involving major muscle groups, performed with body weight or using elastic bands, at moderate to vigorous intensity.
  * Nutrition: will be directed to achieve estimated protein-calorie requirements. Total daily energy requirements will be calculated using the data obtained in the baseline assessment, while daily protein requirements will be set at 1.5 g/kg of body weight. Oral nutritional supplements, particularly a high-calorie, high-protein nutritional blend containing arginine, nucleotides [RNA], and omega-3 fatty acids, will be proposed.
  Arms: Cohort A - neoadiuvant setting - interventional arm
Behavioral: Physical exercise and nutrition for the adjuvant setting — * Physical exercise: 2-3 sessions/week. Each session will be composed of: i) resistance training, including 6-8 exercises for major muscle groups performed in 2-4 sets of 8-12 repetitions; ii) aerobic component, starting at 10-20 minutes, based on the patient's baseline assessments, with monthly progressions up to 40-45 minutes at the end of the program. The insentisy will be set from moderate to vigorous.
  * Nutrition: will be directed to achieve estimated protein-calorie requirements. Total daily energy requirements will be calculated using the data obtained in the baseline assessment, while daily protein requirements will be set at 1.5 g/kg of body weight. Oral nutritional supplements, particularly whey protein, will be proposed.
  Arms: Cohort B - adiuvant setting - interventional arm
Behavioral: Health educational material — Health educational materials, including the benefits of exercise and nutrition during cancer care, the current recommendations and information on how to pursue them, as well as strategies to achieve and maintain a healthy psychological status
  Arms: Cohort B - adiuvant setting

SUMMARY:
The general goal of the STARLighT study is to test whether a structured physical exercise and nutritional intervention significantly impacts clinical outcomes in patients with early-stage lung cancer.

The main questions it aims to answer are:

* Can structured physical exercise and nutrition intervention positively modify the pathological complete response in patients with early-stage lung cancer undergoing neoadjuvant treatments?
* Can structured physical exercise and nutrition intervention positively influence disease-free survival in patients with early-stage lung cancer undergoing adjuvant treatments compared to usual care?

This study will recruit two cohorts of patients. Cohort A will accrue patients who are candidates for neoadjuvant treatment and offer the opportunity to participate in a structured physical exercise and nutritional program, lasting the entire period of anticancer treatment.

Cohort B will accrue patients who are candidates for adjuvant treatments. Patients will be randomized to receive 6 months of structured physical exercise and nutritional intervention or standard of care.

ELIGIBILITY:
Inclusion criteria

* age ≥ 18 years.
* confirmed diagnosis of resectable or resected non-oncogene addicted NSCLC (EGFR, ALK wild-type).
* stage IB to IIIB.
* candidate or undergoing systemic treatment.
* ECOG performance status 0-1.
* written informed consent.
* willingness to use the technology/device specifically developed for patients' monitoring and support within the trial.

Exclusion criteria

* evidence in the medical record of absolute contraindications to exercise, nutritional, or psychological intervention [i.e., heart insufficiency; uncertain arrhythmia; uncontrolled hypertension; severe renal dysfunction, bone marrow insufficiency); reduced standing or walking ability; myocardial infarction].
* indications for or ongoing artificial nutrition support (totally compromised spontaneous food intake).
* incapacity, or unavailability to consume oral nutritional supplements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 324 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2030-04-30 (Estimated); Study Completion 2030-04-30 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response [for Cohort A] | From enrollment up to an average of 3 months
  Defined as a lack of any viable tumor cells after complete evaluation by the local pathologist in the resected lung cancer specimen and all sampled regional lymph nodes.
Quality of life [for Cohort A] | From enrollment up to an average of 3 months
  Assessed using the European Organization for Research and Treatment of Cancer Quality of Life and Core Questionnaire (EORTC QLQ C-30). The scale ranges from 0 to 100; higher values correspond to better quality of life.
Disease-free survival [for Cohort B] | From randomization to the end of follow-up at 2-year.
  Defined as the length of time from study inclusion to recurrence of disease, assessed with the RECIST 1.1 criteria, or death due to any cause.

SECONDARY OUTCOMES:
Treatment toxicities | From enrollment up to 6 months.
  Assessed by the local investigator and categorized according to the Common Terminology Criteria for Adverse Events (version 5.0).
Overall survival | From baseline to the end of follow-up at 2 years.
  Assessed by the local investigator by checking vital status and, eventually, the date of death.
Overall response rate | From enrollment up to 6 months.
  Assessed by the local investigator registering the number of patients who achieve a partial or complete response to the anticancer treatment, according to the RECIST 1.1 criteria.
Disease control rate | From enrollment up to 6 months.
  Assessed by the local investigator registering the number of patients who achieve a stable, partial, or complete response to the anticancer treatment, according to the RECIST 1.1 criteria.
Time to treatment discontinuation | From enrollment up to 6 months.
  Assessed by the local investigator by registering the date and the cause of the treatment discontinuation.
Immuno-inflammatory status | From enrollment up to 6 months.
  Evaluated through the collection of peripheral blood samples. Circulating immuno-inflammatory parameters will be tested using multiplex ELISA.
Functional capacity | From enrollment up to 6 months.
  Assessed with the validated Fitmax Questionnaire, a self-reported questionnaire that estimates cardiorespiratory fitness by quantifying the capacity of walking, cycling, and stair climbing. The scale scores from 0 to 100; higher values correspond to a better functional capacity.
Body mass index | From enrollment up to 6 months.
  Weight and height will be combined to report body mass index in kg/m^2
Muscle mass | From enrollment up to 6 months.
  Estimated using a single-slice transverse CT scan of the third lumbar vertebra, acquired for routine clinical care, using the SliceOmatic version 5.0 (TomoVision) software. This methodology is largely utilized in the oncological setting because it has the advantage of providing high accuracy and reproducible results. The following measure will be quantified: skeletal muscle area (SMA) in cm^2.
Sleep quality | From enrollment up to 6 months.
  Assessed with the Pittsburgh Sleep Quality questionnaire. The scale ranges from 0 to 21. Lower values indicate better sleep quality.
Nutritional risk | From enrollment up to 6 months.
  Assessed with the Nutritional Risk Screening 2002 (NRS-2002). The scale scores from 0 to 7; higher values correspond to a higher risk of malnutrition.
Physical activity level | From enrollment up to 6 months.
  Assessed with the International Physical Activity Questionnaire.
Distress level | From enrollment up to 6 months.
  Assessed with the Distress Thermometer.
Anxiety and Depression levels | From enrollment up to 6 months.
  Assessed with the Hospital Anxiety and Depression Scale. The scale scores from 0 to 42. Higher values correspond to a higher level of anxiety and depression.
Quality of life [for Cohort B] | From enrollment up to 6 months.
  Assessed using the European Organization for Research and Treatment of Cancer Quality of Life and Core Questionnaire (EORTC QLQ C-30). The scale ranges from 0 to 100; higher values correspond to better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Pilotto, Ph.D., MD, Principal Investigator — Universita di Verona
Locations (1):
- Verona Hospital, Verona, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Avancini A, Giannarelli D, Ugel S, Mafficini A, Fiorini P, Scaglione I, Adamoli G, Borsati A, Belluomini L, Eccher S, Trestini I, Tregnago D, Sposito M, Insolda J, Schena F, Scarpa A, Derosa L, Milella M, Novello S, Pilotto S. Telehealth-delivered exercise and nutrition intervention to improve outcomes in patients with early stage non-small cell lung cancer: protocol for the multicentre STARLighT phase II (neoadjuvant) and phase III (adjuvant) trial. BMJ Open. 2026 Jan 12;16(1):e108080. doi: 10.1136/bmjopen-2025-108080. PMID 41526018